CLINICAL TRIAL: NCT00815633
Title: A Pilot Study of Alefacept for the Treatment of Pityriasis Rubra Pilaris.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Failed to enroll patients. There is no data or results for this study.
Sponsor: Joshua Zeichner (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor-Investigator, Joshua Zeichner, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 08-0514; JM-08-001
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Pityriasis Rubra Pilaris
Keywords: PRP; Pityriasis Rubra Pilaris; Amevive; Alefacept; Biologic; Immunosuppressant; Severe skin disease
MeSH Terms: conditions — Pityriasis Rubra Pilaris; Skin Diseases | interventions — Alefacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alefacept (Experimental): Treatment Group (only one group)
  Interventions: Drug: Alefacept

INTERVENTIONS:
Drug: Alefacept — 15mg intramuscular injection weekly for 12 weeks
  Other Names: Amevive

SUMMARY:
The purpose of this study is to determine whether the biologic medication alefacept (Amevive) is effective and safe in the treatment of Pityriasis Rubra Pilaris.

DETAILED DESCRIPTION:
Pityriasis Rubra Pilaris (PRP) is a therapeutic challenge, and many different medication regimens exist to treat the condition. Clinical response is variable, and no single treatment has emerged as a leading therapy. Biologic agents have emerged as effective treatments for many skin diseases, including psoriasis. Given the clinical overlap between PRP and psoriasis, it is logical to attempt to use these agents for PRP. Since the majority of patients with PRP are unresponsive to current therapies, new treatment modalities must be evaluated. This study will evaluate the treatment of adult 30 years or older with a diagnosis of PRP, either subtypes 1 or 2. In this study, the safety and efficacy of alefacept will be evaluated in adult patients with PRP refractory to current treatments. Alefacept is a dimeric fusion protein containing the CD2 extracellular binding region of human leukocyte function antigen-3 (LFA-3) linked to the Fc portion of human IgG1. The drug binds to the T-lymphocyte antigen CD2 and blocks its interaction with LFA-3 on antigen presenting cells in the body. The CD2/LFA-3 interaction is a key co-stimulatory signal in the activation of T-lymphocytes central to the pathophysiology of psoriasis. It is theorized this interaction plays a role in the pathophysiology of PRP. Alefacept is currently approved for the treatment of adults with moderate to severe, chronic, plaque-type psoriasis. The medication is administered as weekly intramuscular injections for 12 week courses. In this study, a dose of 15mg alefacept will be administered intramuscularly at weekly intervals for 12 weeks. This is the dosing regimen currently approved for the treatment of psoriasis. Patients will be followed for a total of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be male or female, 30 years old or older at time of consent
* Have a diagnosis of pityriasis rubra pilaris at least 6 months prior to administration of the first dose of the study medication
* Be a candidate for systemic therapy
* Women of childbearing potential and all men must use adequate contraceptive measures if sexually active. Examples include abstinence, oral contraceptives or other form of hormonal contraception, intrauterine devices, surgical sterilization, or barrier forms of contraception with spermicidal jelly. Subjects must agree to continue to use these contraceptive measures and agree not to become or plan a pregnancy within 12 months of the date of the last study drug administration.
* Agree to adhere to the study visit schedule and protocol requirements, including blood draws and clinical photographs.
* Must be able to give informed consent, and this consent must be obtained prior to any study related procedures being performed.
* Must avoid other treatment modalities during the course of the study and adhere to standard washout periods for any medications used to treat their skin prior to receiving the first dose of study medication.
* Must agree not to receive a live viral or bacterial vaccine during the course of the study or for 12 months after the date of the last study drug administration.
* Have screening blood tests that are stable as deemed by the physician investigator. AST, ALT and alkaline phosphatase levels must be within 2.0 times the upper limit of normal to participate.

Exclusion Criteria:

* Subjects are pregnant or planning a pregnancy (both men and women) while enrolled in the study.
* Have used the medication alefacept in the past.
* Have used another investigational medication within the past 4 weeks or within 5 times the half-life of that investigational medicine.
* Have received systemic medications that could affect pityriasis rubra pilaris within 4 weeks of administration of the first dose of the study medicine.
* Have used topical medications that could affect pityriasis rubra pilaris within 2 weeks of administration of the first dose of the study medicine.
* Have received a live viral or bacterial vaccine within 3 months of administration of the first dose of the study medicine.
* Have a history of chronic or recurrent infections of the skin or internal organs.
* Have had a serious infection requiring hospitalization or intravenous antibiotics within 2 weeks of administration of the first dose of the study medicine.
* Have a history of latent untreated tuberculosis.
* Have a known history of human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus.
* Have a history of a malignancy except for squamous cell or basal cell carcinoma of the skin or cervical carcinoma in situ that has been treated with no evidence of recurrence.
* Have a known hypersensitivity to any component of alefacept.
* Have a known substance abuse problem or is deemed by the investigator as unable to follow the study protocol.
* Is participating in another study for an investigational agent or procedure during the course of this study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Zeichner, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alefacept
Started | 1
Completed | 0
Not Completed | 1
Not completed — study terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Alefacept
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Skin Change - Physician's Global Assessment (PGA)
Time Frame: wks 1,2,3,4,5,6,7,8,9,10,11,12, 16,20,24
Population: study terminated before data collected
Arm/Group | Alefacept
Number analyzed (Participants) | 0

2. Primary Outcome: Evidence of Skin Change - PRP Area and Severity Index (PASI)
Time Frame: wks 1,2,3,4,5,6,7,8,9,10,11,12, 16,20,24
Population: study terminated before data collected
Arm/Group | Alefacept
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: adverse events not collected
Arm/Group | Alefacept
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes